CLINICAL TRIAL: NCT05771896
Title: A Phase III Randomized Study Comparing the Combination of Darolutamide With Radium-223 or Placebo and the Effect on Radiological Progression-Free Survival for Patients With Metastatic Castration-Sensitive Prostrate Cancer (mCSPC)
Brief Title: Darolutamide With Radium-223 or Placebo and the Effect on Radiological Progression-Free Survival for Patients With mCSPC
Acronym: CARE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Bayer withdrew their support.
Sponsor: GenesisCare USA (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00019_CARE
Record Dates: First submitted 2023-02-06; First posted 2023-03-16 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Radium-223; radium Ra 223 dichloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Darolutamide with Radium-223 (Experimental): Darolutamide:
  Dosage:600mg Route: By mouth (PO) Frequency: Twice a day, throughout the duration of the study
  Radium-223:
  Dosage: 55 kBq/kg body weight or 1.49 microcurie/kg body weight Route: IV Frequency: Every 28+/-7 days, a maximum of 6 cycles
  Interventions: Drug: Darolutamide; Drug: Radium-223
- Darolutamide with Placebo (Placebo Comparator): Darolutamide:
  Dosage:600mg Route: By mouth (PO) Frequency: Twice a day, throughout the duration of the study
  Placebo:
  Dosage: 55 kBq/kg body weight or 1.49 microcurie/kg body weight Route: IV Frequency: Every 28+/-7 days, a maximum of 6 cycles
  Interventions: Drug: Darolutamide

INTERVENTIONS:
Drug: Darolutamide — Participants will continue treatment with darolutamide until radiological progression, withdrawal, death, termination, or study completion.
  The maximum time for darolutamide dose interruption period is 28 consecutive days beyond scheduled dose (>56 days between cycles). Any participant requiring dose interruption >28 consecutive days beyond the scheduled dose may restart treatment with darolutamide if clinical benefit is anticipated and after discussion with and approval from the study Medical Monitor.
  Until primary endpoint is reached, participants are not allowed to switch ARPI (Abiraterone, Apalutamide or Enzalutamide) during the study. Switching to other ARPI following radiographic progression should be considered a subsequent life prolonging therapy and documented accordingly.
  Other Names: Nubeqa
Drug: Radium-223 — Radium-223 should be given for 6 cycles, administered IV on Day 1 of each cycle or until radiological progression, withdrawal, death, termination, or study completion. The placebo will be administered in precisely the same fashion as the active drug.
  Subsequent cycles 2-6 should be scheduled to occur every 28 ± 7 days following the previous cycle, but dosing may be delayed up to 28 days per cycle (maximum 56 days between cycles). Any participant requiring dose interruption >28 consecutive days (>56 days between cycles) may restart treatment with radium-223/placebo if clinical benefit is anticipated and after discussion with the Medical Monitor. Participants will continue with darolutamide irrespective of Radium-223 administration.
  Upon radiological progression, further treatments are decided by the site investigator according to standard local practice.
  Other Names: Xofigo
  Arms: Darolutamide with Radium-223

SUMMARY:
The goal of this clinical trial is to compare the combination of Darolutamide with Radium-223 or placebo and the effects on radiological progression-free survival for patients with Metastatic Castration-Sensitive Prostrate Cancer (mCSPC)

The main questions it aims to answer are:

* Radiological progression-free survival (rPFS) in mCSPC
* Overall Survival (OS)
* Symptomatic skeletal event-free survival (SSE-FS)
* Initiation of subsequent antineoplastic therapy
* Safety

Participants will have visits at baseline, treatment is once a month for up to 6 months, and long term follow up will continue until the participant dies, withdraws consent, and/or study is terminated.

DETAILED DESCRIPTION:
A novel treatment strategy combining darolutamide and radium-223 is considered for subjects with mCSPC. Response to treatment is monitored every 12 weeks using a continuous measurement. The main scientific question concerns the comparison of radium-223 to placebo and is best addressed by a randomized clinical trial. Use of placebo in this study is considered ethical, as provision is made for subjects to discontinue their treatment and switch to radium-223 due to lack of efficacy on unblinding where it influences current treatment decisions. Switch to rescue medication is an intercurrent event, after which it is still possible to collect the variable measurements as described in sections on study endpoints below. This is also the case after other intercurrent events such as discontinuation of radium-223 treatment due to an adverse event, but not for intercurrent events such as death unrelated to study IP or disease, subject loss to follow-up, or subject withdrawal from all study treatments and procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able and willing to provide informed consent.
2. Metastatic castration-sensitive prostate cancer (mCSPC) at screening with histologically or cytologically confirmed diagnosis of prostate adenocarcinoma.
3. Men ≥ 18 years.
4. ECOG performance status of 0, 1 or 2 at screening.
5. Metastatic to bone with ≥ 2 bone metastases (area of increased uptake on 99mTc methylene diphosphonate bone scan); equivocal lesions on the bone scan must be confirmed by standard X-ray, CT, or MRI.
6. Ongoing ADT by Investigator's choice with luteinizing hormone-releasing hormone (LHRH) agonist or antagonist or bilateral orchiectomy for less than 120 days prior to randomization. ADT treatment should be on a stable dose without interruptions of at least 4 weeks prior to first dose of blinded IP.
7. On bone health agents with at least one dose of BHA prior to first dose of blinded IP.
8. Adequate bone marrow and organ function as defined by:

   1. Hemoglobin ≥ 9.0 g/dL
   2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   3. Platelets ≥ 100 x 109/L (participant must not have received any growth factor within 4 weeks or a blood transfusion within 7 days of the hematology laboratory sample obtained at Screening)
   4. Serum creatinine ≤2 x upper limit of normal ULN
   5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 1.5 x upper limit of normal (ULN)
   6. Total bilirubin < 1.5 x ULN, unless the participant a diagnosis of Gilbert's disease or a similar syndrome involving slow conjugation of bilirubin; in participants with Gilbert's, the total bilirubin should be < 3 x ULN and the elevation should be seen in the unconjugated or indirect bilirubin measurement)
   7. Albumin ≥ 2.5 g/dL
9. Fertile male participants, defined as all males physiologically capable of conceiving offspring with female partners of child-bearing potential, must be willing to use condoms plus spermicidal agent during the study treatment period and for 6 months after the last dose of blinded IP, and not father a child or donate sperm during this period.
10. No known contraindication to any study treatment (darolutamide, radium-223, and/or Investigator's choice ADT).

Exclusion Criteria:

1. Pathological finding consistent with small cell carcinoma of the prostate.
2. Prior treatment for mCSPC [excluding ADT ≤120 days and first-generation ARI (bicalutamide, nilutamide or flutamide) for ≤120 days when initiating ADT], with the exception of Metastases Directed Therapy (MDT) with EBRT/SBRT (at least 2 bone metastases must be untreated). Prior treatment for localized prostate cancer is allowed (all treatments must have been completed ≥ 1 year prior to randomization)
3. Treatment for mCSPC with ADT starting >120 days prior to randomization.
4. Treatment for mCSPC with first generation ARI (bicalutamide, nilutamide or flutamide) starting >120 days prior to randomization.
5. Prior hemi-body or whole-body external radiotherapy.

   a. Other types of prior external radiotherapy and brachytherapies are allowed, if more than 28 days prior to randomization.
6. Prior therapy with radionuclides (e.g., including but not limited to radium-223, strontium-89, samarium-153), including prior therapy with investigational radionuclides (e.g., including but not limited to iodine-131, rhenium-186, rhenium- 188, thorium- 277, actinium-225 and lutetium-177).
7. Prior treatment with:

   * Second-generation androgen receptor (AR) inhibitors such as enzalutamide, darolutamide, apalutamide or other investigational AR inhibitors.
   * Cytochrome P 17 enzyme inhibitor such as abiraterone acetate or oral ketoconazole as antineoplastic treatment for prostate cancer.
   * Chemotherapy including docetaxel or immunotherapy for prostate cancer.
   * Use of systemic corticosteroid with dose greater than the equivalent 10 mg of prednisone/day within 28 days prior to randomization.
8. Current involvement in any drug or device trial involving investigational agent or medical device within the last 28 days prior to randomization.
9. Any prior investigational agent for nmCSPC/mCSPC.
10. Known hypersensitivity to compounds related to darolutamide, or radium-223, or to CT and/or MRI contrast media.
11. A blood transfusion ≤ 28 days prior to randomization.
12. Major surgical procedures ≤ 28 days or minor surgical procedures ≤7 days prior to randomization. No waiting period is required following port-a-cath placement.
13. Superscan on 99mTc methylene diphosphonate bone scan.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with Metastatic Castration-Sensitive Prostrate Cancer
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Radiological progression-free survival (rPFS) in mCSPC patients | First occurrence bone scan progression and/or soft tissue progression per #RECIST 1.1 criteria, participant dies, withdraws consent and/or study is terminated, whichever comes first.
  The primary objective of this study is to compare the radiological progression-free survival (rPFS) in mCSPC patients treated with darolutamide plus radium-223 versus darolutamide plus placebo. The primary endpoint is radiological progression-free survival rPFS, defined as time to first occurrence of 99mTc MDP+ bone scan progression per PCWG3 criteria, and/or soft tissue progression by CT/MRI per PCWG3 modifications to RECIST 1.1 criteria, or death from any cause. Randomization will be stratified by ECOG performance status 0 vs 1-2, and metastatic disease status, specifically low volume (<4 bone lesions) versus high volume (≥4 bone lesions).

SECONDARY OUTCOMES:
Overall Survival (OS) & Symptomatic Skeletal Event-Free Survival (SSE-FS) | Randomization until death.
  Overall survival and SSE-FS will be compared between the two arms using a stratified log-rank test, HR (Darolutamide + radium-223 dichloride / Darolutamide + placebo) with 95% CI. Kaplan-Meier estimates and plots for both treatment arms will be produced to accompany these analyses. The median, 25th and 75th percentiles and event free rates at different timepoints with associated 95% CI will be generated.
  SSE-FS as defined as the time from randomization until any one of the following:
  * the first use of external-beam radiation therapy to relieve skeletal tumor-related symptoms,
  * the occurrence of new symptomatic pathologic bone fractures,
  * the occurrence of new symptomatic spinal cord compression,
  * a tumor-related orthopedic surgical intervention, or
  * death.
Initiation of Subsequent Antineoplastic Therapy | Randomization to initiation of first subsequent antineoplastic therapy for prostrate cancer.
  Time to initiation of subsequent antineoplastic therapy will be compared considering death as a competing risk. Treatment arms will be compared with stratified competing risk HR (Darolutamide + radium-223 dichloride / Darolutamide + placebo) with 95% CI. Event rates will be estimated by cumulative incidence.
Safety of the combination of radium-223 and Darolutamide | First treatment dose until last dose + 30 Days
  Safety of the combination of radium-223 and Darolutamide will be assessed by the incidence, nature, and severity of adverse events (AEs) and serious adverse events (SAEs) per Common Toxicity Criteria for Adverse Events (CTCAE) v5.0. Exposure-adjusted incidence rates (EAIR) may be provided.

IPD SHARING:
Plan to Share IPD: No